CLINICAL TRIAL: NCT03344393
Title: Effect of Intraoperative IV Ketamine on Postoperative Morphine Consumption During Intestinal Surgery and Its Effect on Salivary Cortisol and Alpha Amylase Levels
Brief Title: Effect of Intraoperative IV Ketamine on Postoperative Morphine Consumption During Intestinal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed galal aly, Assistant Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17200147
Record Dates: First submitted 2017-11-09; First posted 2017-11-17 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Postoperative Analgesia
MeSH Terms: interventions — Ketamine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ketamine hydrochloride (Active Comparator): intravenous ketamine infusion in the intraoperative period
  Interventions: Drug: Ketamine Hydrochloride
- normal saline (Active Comparator): intravenous normal saline infusion in the intraoperative period
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ketamine Hydrochloride — intravenous ketamine infusion intraoperatively
  Other Names: ketalar
  Arms: ketamine hydrochloride
Drug: Normal saline — intravenous normal saline infusion intraoperatively
  Other Names: Sodium chloride solution
  Arms: normal saline

SUMMARY:
.The aim of this study is to identify the analgesic effect of intraoperative ketamine intravenous infusion on patients undergoing intestinal surgery and its effect on salivary cortisol and alpha amylase levels as indicator of its effect.

DETAILED DESCRIPTION:
I- Group K (ketamine): 30 patients will receive intraoperative intravenous ketamine infusion.

II- Group C (control): 30 patients will receive intraoperative intravenous normal saline infusion.

ELIGIBILITY:
Inclusion Criteria:

* - Patient's status ASA status-I and II.
* Patients age above 18 years old.
* Patients scheduled for intestinal surgery.

Exclusion Criteria:

* Patient refusal.
* Patients with known allergy to ketamine or morphine.
* Patients with significant hepatic dysfunction.
* Patients with severe renal disease.
* Significant Heart disease.
* Patients with chronic pain.
* Regular use analgesics, antidepressants or opioids in last 2 months.
* Any known convulsive disorder.
* Morbid obesity (BMI>35).
* Patients with autoimmune disease
* Patients on corticosteroid therapy
* Pregnancy.
* Breast feeding.
* Woman under hormonal treatment.
* Oral disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — above 18
Enrollment: 60 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
morphine consumption | 2 days postoperative
  IV PCA

SECONDARY OUTCOMES:
cortisol level | 2 days postoperative
  salivary
alpha amylase level | 2 days postoperative
  salivary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arikan M, Aslan B, Arikan O, Horasanli E, But A. Comparison of the effects of magnesium and ketamine on postoperative pain and morphine consumption. A double-blind randomized controlled clinical study. Acta Cir Bras. 2016 Jan;31(1):67-73. doi: 10.1590/S0102-865020160010000010. PMID 26840358